CLINICAL TRIAL: NCT02723331
Title: Perioperative Therapy for Resectable Pancreatic Adenocarcinoma and Borderline Resectable Pancreatic Adenocarcinoma With Molecular Correlates
Brief Title: Perioperative Therapy for Resectable and Borderline-Resectable Pancreatic Adenocarcinoma With Molecular Correlates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic Thoracic Oncology Medical Investigators Consortium (Industry)
Collaborators: Celgene Corporation (Industry); Criterium, Inc. (Industry); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Organization: University of Colorado, Denver (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0150.cc
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreas Ductal Adenocarcinoma
Keywords: Stereotactic Body Radiation Therapy; Perioperative Therapy; Resectable Pancreas Ductal Adenocarcinoma; Borderline Resectable Pancreas Ductal Adenocarcinoma; Nab-paclitaxel; Abraxane; Gemcitabine; Neoadjuvant Therapy; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nab-paclitaxel and Gemcitabine for R-PDAC (Experimental): Nab-paclitaxel and gemcitabine, for R-PDAC patients enrolled in this trial, will be given in combination as neoadjuvant combination chemotherapy, followed by SBRT. This is will be followed up by surgical resection and an additional combination chemotherapy of nab-paclitaxel and gemcitabine as adjuvant chemotherapy.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine
- Nab-paclitaxel and Gemcitabine for BR-PDAC (Experimental): Nab-paclitaxel and gemcitabine, for BR-PDAC patients enrolled in this trial, will be given in combination as neoadjuvant combination chemotherapy, followed by SBRT. This is will be followed up by surgical resection and an additional combination chemotherapy of nab-paclitaxel and gemcitabine as adjuvant chemotherapy.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab paclitaxel — Nab-paclitaxel and gemcitabine, for R-PDAC patients, will be given in combination as neoadjuvant and adjuvant chemotherapy. Nab-paclitaxel will be administered by IV infusion at a dose of 125 mg/m2 over 30 minutes on Days 1, 8, and 15 of every 28-day cycle. Gemcitabine will be administered by IV infusion, immediately after the administration of nab-paclitaxel, at a dose of 1000 mg/m2 over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Other Names: Abraxane
Drug: Gemcitabine — Nab-paclitaxel and gemcitabine, for BR-PDAC patients, will be given in combination as neoadjuvant and adjuvant chemotherapy. Nab-paclitaxel will be administered by IV infusion at a dose of 125 mg/m2 over 30 minutes on Days 1, 8, and 15 of every 28-day cycle. Gemcitabine will be administered by IV infusion, immediately after the administration of nab-paclitaxel, at a dose of 1000 mg/m2 over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
  Other Names: Gemzar

SUMMARY:
The objective of this study is to estimate the R0 resection rate in patients with Resectable Pancreatic Ductal Adenocarcinoma (R-PDAC) as well as those with Resectable Pancreatic Ductal Adenocarcinoma (BR-PDAC) independently in response to neoadjuvant sequential therapy of combination nab-paclitaxel and gemcitabine followed by stereotactic body radiotherapy (SBRT).

DETAILED DESCRIPTION:
Patients in both cohorts will receive a total of 3 cycles of neoadjuvant combination chemotherapy of nab-paclitaxel and gemcitabine, followed by re-staging CT scan, if re-staging CT does not show evidence of metastatic disease. Patients will receive SBRT and definitive surgical resection. Subsequently, patients will receive 3 cycles of adjuvant combination chemotherapy of nab-paclitaxel and gemcitabine. Each cycle of combination chemotherapy will be a total of 4 weeks. Patients will be evaluated for response at completion of the 3 cycles of neoadjuvant combination chemotherapy with CT scans of chest, abdomen and pelvis. Patients will undergo surveillance CT scan at 3-month intervals until evidence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed resectable or borderline resectable pancreatic adenocarcinoma.
2. No evidence of distant metastasis representing stage IV metastatic disease.
3. R-PDAC: No evidence of distant metastasis and tumor mass showing no extension to superior mesenteric artery (SMA) and hepatic artery. There must be a clearly defined fat plane between SMA and celiac axis. Patent superior mesenteric vein (SMV/portal vein (PV) with no distortion of venous architecture.
4. BR-PDAC: defined as localized PDAC with 1 or more of the following features: a) an interface between the primary tumor and superior mesenteric vein (SMV)-portal vein (PV) measuring 180o or greater of the circumference of the vein wall, and/or b) short-segment occlusion of the SMV-PV with normal vein above and below the level of obstruction that is amenable to resection and venous reconstruction and/or c) short-segment interface of any degree between tumor and hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and arterial reconstruction and/or d) an interface between the tumor and SMA or celiac trunk measuring less than 180o of the circumference of the artery wall.
5. Age > 18 years old
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Patients must have adequate bone marrow function:

   * Platelets >100,000 cells/mm3
   * Hemoglobin > 9.0 g/dL
   * Absolute Neutrophil Count > 1,500 cells/mm3
8. Patients must have adequate liver function:

   * aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2.5 X upper limit of normal
   * Alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
   * Total bilirubin < 1.5 mg/dL
9. Patients must have adequate renal function: creatinine <1.5 mg/dL is recommended; however, institutional norms are acceptable. Creatinine within institutional limits of normal or creatinine clearance (CrCl) > 50 mL/min calculated using the Cockcroft-Gault equation.
10. Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment.
11. Negative serum or urine β-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of childbearing potential.
12. Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE 4.03).
13. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients with locally advanced surgically unresectable PDAC.
2. Patients with evidence of distant metastatic PDAC.
3. Prior chemotherapy or radiation therapy of any kind for treatment of pancreas adenocarcinoma.
4. Prior major surgery within 4 weeks of starting study drug administration.
5. Patient unable or not willing to perform all study related biopsies and blood draws for exploratory endpoints will not be enrolled on study as all study related procedures are mandatory.
6. Concomitant treatment with full dose warfarin (coumadin) is NOT allowed. However, treatment with low molecular weight heparin (LMWH) (such as enoxaparin or dalteparin) or rivaroxaban is allowed. Patients on full dose warfarin (coumadin) must be transitioned to either LMWH or rivaroxaban prior to administration of any study related drugs.
7. Recent or ongoing clinically significant gastrointestinal disorder (e.g., malabsorption, bleeding, inflammation, emesis, diarrhea >grade 1).
8. Patients with clinically significant cardiac disease (New York Heart Association Classification III or IV and cardiac arrhythmias not well controlled with medication), or myocardial infarction within the previous six months.
9. Serious, uncontrolled, concurrent infection(s) requiring antibiotics.
10. Pregnant or breastfeeding women: positive pregnancy test within 7 days of starting treatment.
11. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
12. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
13. Patients with external biliary drains.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen DJ, Goldberg JD, Leichman L, Hochman T, Newman E, Du K, Megibow A, Oberstein P, Al-Rajabi R, Scott AJ, Bekaii-Saab T, Messersmith WA, Weekes C. Perioperative therapy for resectable and borderline resectable pancreatic adenocarcinoma: an Academic Gastrointestinal Cancer Consortium Study. Oncologist. 2025 Oct 1;30(10):oyaf271. doi: 10.1093/oncolo/oyaf271. PMID 40972532

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-paclitaxel/Gemcitabine for R-PDAC: Nab-paclitaxel and gemcitabine, for R-PDAC patients enrolled in this trial, will be given in combination as neoadjuvant combination chemotherapy, followed by SBRT. This is will be followed up by surgical resection and an additional combination chemotherapy of nab-paclitaxel and gemcitabine as adjuvant chemotherapy.
  Nab-paclitaxel and gemcitabine for R-PDAC Patients: Nab-paclitaxel and gemcitabine, for R-PDAC patients, will be given in combination as neoadjuvant and adjuvant chemotherapy. Nab-paclitaxel will be administered by IV infusion at a dose of 125 mg/m2 over 30 minutes on Days 1, 8, and 15 of every 28-day cycle. Gemcitabine will be administered by IV infusion, immediately after the administration of nab-paclitaxel, at a dose of 1000 mg/m2 over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
- Nab-paclitaxel/Gemcitabine for BR-PDAC: Nab-paclitaxel and gemcitabine, for BR-PDAC patients enrolled in this trial, will be given in combination as neoadjuvant combination chemotherapy, followed by SBRT. This is will be followed up by surgical resection and an additional combination chemotherapy of nab-paclitaxel and gemcitabine as adjuvant chemotherapy.
  Nab-paclitaxel and gemcitabine for BR-PDAC Patients: Nab-paclitaxel and gemcitabine, for BR-PDAC patients, will be given in combination as neoadjuvant and adjuvant chemotherapy. Nab-paclitaxel will be administered by IV infusion at a dose of 125 mg/m2 over 30 minutes on Days 1, 8, and 15 of every 28-day cycle. Gemcitabine will be administered by IV infusion, immediately after the administration of nab-paclitaxel, at a dose of 1000 mg/m2 over 30 minutes on Days 1, 8 and 15 of every 28-day cycle.
Period: Overall Study
Arm/Group | Nab-paclitaxel/Gemcitabine for R-PDAC | Nab-paclitaxel/Gemcitabine for BR-PDAC
Started | 19 | 29
Completed | 3 | 5
Not Completed | 16 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-paclitaxel and Gemcitabine for R-PDAC | Nab-paclitaxel and Gemcitabine for BR-PDAC | Total
Number analyzed (Participants) | 19 | 29 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.35 (8.3) | 68.4 (8.8) | 68.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 15 | 26 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 3 | 3
  White | 16 | 24 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 19 | 29 | 48

OUTCOME MEASURES:

1. Primary Outcome: R0 Resection Rates in Each Cohort as Measured by Macroscopically Complete Tumor Removal With Negative Microscopic Surgical Margins
Description: R0 resection rates will be measured in patients with resectable PDAC and with patients with borderline-resectable PDAC, independently in response to neoadjuvant sequential therapy of combination of nab-paclitaxel and gemcitabine and SBRT, as perioperative therapy. R0 resection is determined by macroscopically complete tumor removal with negative microscopic surgical margins in the bile duct, pancreatic parenchyma, and superior mesenteric artery (SMA).
Time Frame: at the time of surgery
Measure: Number; unit: participants with resectable PDAC
Arm/Group | Nab-paclitaxel/Gemcitabine for R-PDAC | Nab-paclitaxel/Gemcitabine for BR-PDAC
Number analyzed (Participants) | 19 | 29
participants with resectable PDAC | 9 | 9

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v.4.03
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel/Gemcitabine for R-PDAC | Nab-paclitaxel/Gemcitabine for BR-PDAC
Number analyzed (Participants) | 19 | 29
Participants | 19 | 29

3. Secondary Outcome: Median Overall Survival
Description: Overall survival will be assessed for all participants
Time Frame: Up to 74 months
Measure: Median (Full Range); unit: months
Arm/Group | Nab-paclitaxel/Gemcitabine for R-PDAC | Nab-paclitaxel/Gemcitabine for BR-PDAC
Number analyzed (Participants) | 19 | 29
months | 17.4 [5.2 to 53.6] | 15.5 [1 to 73.7]

ADVERSE EVENTS:
Time Frame: Up to 74 months
Arm/Group | Nab-paclitaxel/Gemcitabine for R-PDAC | Nab-paclitaxel/Gemcitabine for BR-PDAC
All-Cause Mortality (participants affected / at risk) | 18/19 | 26/29
Serious Adverse Events (participants affected / at risk) | 10/19 | 17/29
Other Adverse Events (participants affected / at risk) | 19/19 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel/Gemcitabine for R-PDAC (N=19) | Nab-paclitaxel/Gemcitabine for BR-PDAC (N=29)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Biliary Obstruction (Hepatobiliary disorders) | 2 (2) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (3)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Failure to Thrive (General disorders) | 1 (1) | 0 (0)
GI infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Creatinine (Investigations) | 1 (1) | 0 (0)
Gastric Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Renal Calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Duodenal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Uncontrolled Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ischemic Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jaundice (Investigations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bleeding (post operative) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SIRS (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel/Gemcitabine for R-PDAC (N=19) | Nab-paclitaxel/Gemcitabine for BR-PDAC (N=29)
Abdominal Cramps (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Distention / Bloating (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 12 (15) | 11 (17)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 3 (5) | 5 (12)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7) | 10 (10)
Alanine Aminotransferase increased (Investigations) | 7 (10) | 5 (11)
Anal Hemorrhage (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 13 (43) | 18 (43)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Anisocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorectal pain (General disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 7 (7)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 7 (15) | 7 (17)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 2 (2) | 3 (4)
Bilateral edema (Blood and lymphatic system disorders) | 4 (7) | 11 (11)
Biliary Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 3 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Chest wall pain (Cardiac disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 6 (6) | 3 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Clostridium difficile colitis (Investigations) | 1 (1) | 0 (0)
confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (14) | 14 (15)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3)
Creatinine Increased (Investigations) | 2 (3) | 4 (7)
Activity change (General disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (7) | 6 (12)
Thrombocytopenia (Investigations) | 5 (10) | 8 (16)
Leukopenia (Investigations) | 9 (19) | 11 (24)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (16) | 13 (15)
Dizziness (Nervous system disorders) | 3 (5) | 5 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (5) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (8)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Epistaxis (General disorders) | 4 (4) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Fatigue (General disorders) | 16 (25) | 22 (30)
Fever (General disorders) | 8 (11) | 8 (10)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Flu like Symptoms (Investigations) | 3 (3) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 3 (3)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Headache (General disorders) | 5 (5) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (14) | 6 (12)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (10) | 7 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8) | 3 (5)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 6 (6)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 4 (8) | 8 (12)
Mucositis Oral (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 13 (16) | 16 (21)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Neuropathy (Nervous system disorders) | 9 (13) | 12 (14)
Neutropenia (Blood and lymphatic system disorders) | 11 (19) | 20 (42)
Pain (general) (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (11)
Pancreatic Insufficiency (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 5 (6)
Rash (general) (Skin and subcutaneous tissue disorders) | 6 (9) | 6 (13)
Sore Throat (Gastrointestinal disorders) | 0 (0) | 3 (4)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (9) | 9 (13)
Weight Loss (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Concentration Impairment (General disorders) | 1 (1) | 0 (0)
Decreased Absolute Monocytes (Investigations) | 1 (1) | 1 (1)
Decreased Urine Volume (Renal and urinary disorders) | 1 (1) | 0 (0)
Difficulty Urinating (Renal and urinary disorders) | 1 (1) | 0 (0)
Distended loops of bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
dysuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Emboli (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Transaminitis (Investigations) | 1 (1) | 1 (1)
Tremor (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Venous Thrombosis (Vascular disorders) | 1 (1) | 2 (3)
Elevated INR (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nail Discooeration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT02723331/Prot_SAP_ICF_000.pdf